CLINICAL TRIAL: NCT04858126
Title: Accuracy of the ECOM Plus Hemodynamic Monitor Versus Pulmonary Artery Catheter
Brief Title: Accuracy of ECOM Plus Versus Pulmonary Artery Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECOM Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECOM SP 20-007
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-01

CONDITIONS: Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Group Assignment (Experimental): ECOM endotracheal cardiac output monitor in patients undergoing cardiac and liver surgery.
  Interventions: Device: ECOM cardiac output

INTERVENTIONS:
Device: ECOM cardiac output — Measure cardiac output during perioperative period and compare to pulmonary artery catheter thermal dilution cardiac output measurement.

SUMMARY:
This Study will compare the accuracy of the ECOM Plus Endotracheal Cardiac Output Monitor (ECOM) without the use of the arterial pressure waveform from the arterial line to 1) the current clinical standard of cardiac output measured by intermittent room temperature bolus thermodilution using a PAC, 2) the current ECOM System with the use of the arterial blood pressure waveform from a radial arterial line and 3) the Flo-Trac® System.

DETAILED DESCRIPTION:
This Study will compare the accuracy of the ECOM Plus Endotracheal Cardiac Output Monitor (ECOM) without the use of the arterial pressure waveform from the arterial line to 1) the current clinical standard of cardiac output measured by intermittent room temperature bolus thermodilution using a PAC, 2) the current ECOM System with the use of the arterial blood pressure waveform from a radial arterial line and 3) the Flo-Trac® System (Edwards LifeSciences).

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed consent.
* Patients undergoing surgery that would routinely require use of an endotracheal, pulmonary artery catheter and arterial catheter.

Exclusion Criteria:

* Patients who do not speak English.
* Patients not competent to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Comparison of ECOM Plus impedance and thermal dilution cardiac output measurements | 6 months.
  Correlation via linear regression between thermal dilution and ECOM Plus included as an "R" to coefficient. Cardiac output measured by thermal dilution and impedance cardiography. Management of the patients using standard thermal dilution derived CO measurement only. The ECOM Plus measurement output are for research purposes only and not to be used in the management of the patient. ECOM Plus impedance cardiography measured in the ICU when routine thermal dilution CO measurements are made. Continued impedance measurements until tracheal extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wallace, MD, Principal Investigator — VA San Francisco
Locations (1):
- VA San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Data and information for 510(k).

REFERENCES:
- [Background] Wallace AW, Salahieh A, Lawrence A, Spector K, Owens C, Alonso D. Endotracheal cardiac output monitor. Anesthesiology. 2000 Jan;92(1):178-89. doi: 10.1097/00000542-200001000-00030. PMID 10638915